CLINICAL TRIAL: NCT06875973
Title: A Rollover Extension Program (REP) to Evaluate the Long-term Safety and Tolerability of Open-Label Pelacarsen in Participants With Elevated Lp(a) and Established ASCVD
Brief Title: Pelacarsen Roll-over Extension Program
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTQJ230A12305B
Record Dates: First submitted 2025-03-12; First posted 2025-03-14 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Atherosclerotic Cardiovascular Disease
Keywords: TQJ230; Lp(a); ASCVD
MeSH Terms: conditions — Atherosclerosis | interventions — pelacarsen

STUDY DESIGN:
Intervention Model Description: Rollover extension program (REP)
Masking Description: Open label study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pelacarsen (TQJ230) (Experimental): open-label pelacarsen 80mg
  Interventions: Drug: Pelacarsen (TQJ230)

INTERVENTIONS:
Drug: Pelacarsen (TQJ230) — pelacarsen 80mg s.c. monthly
  Other Names: TQJ230

SUMMARY:
This non-randomized, rollover extension study will provide post-trial access to pelacarsen (TQJ230) to participants who have successfully completed either of the double-blind parent studies (CTQJ230A12303 or CTQJ230A12304).

DETAILED DESCRIPTION:
This study will evaluate long-term safety and tolerability of pelacarsen (TQJ230) 80 mg Once a month (QM) in patients with elevated Lp(a) and established ASCVD. All consenting participants from the parent study who meet the eligibility criteria will be participating in this open label extension study.

ELIGIBILITY:
Inclusion Criteria:

* Participants who have provided informed consent prior to initiation of any study-specific activities/procedures.
* Participants who have completed the parent study and received the assigned study treatment at the time of its completion

Exclusion Criteria:

* Participants who permanently discontinued the study treatment as mandated per protocol or due to adverse events in the parent study
* Any medical condition(s) in the investigator's opinion that may put the participant at risk or interfere with the study participation
* Participants who are receiving another investigational drug or device before the open-label treatment period
* Participants who have a known sensitivity to the study drug and are deemed as unsuited for the study by the investigator

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2025-05-19 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-01-03 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse events (AEs) or serious adverse events (SAEs) | 36 months
  Evaluate long-term safety and tolerability of pelacarsen (TQJ230) in participants with elevated Lp(a) and established atherosclerotic cardiovascular disease who have completed the parent study

SECONDARY OUTCOMES:
Observed value and change in Lipoprotein(a) (Lp(a)) compared to baseline of the parent study | Baseline of the core study, Month 3, 12, 24, 36, 48
  Evaluate the long-term efficacy of pelacarsen (TQJ230) in lowering Lp(a) levels
Observed value and change in Lp(a) compared to baseline of the rollover extension program (REP) study | Baseline of the REP study, Month 3, 12, 24, 36, 48
  Evaluate the long-term efficacy of pelacarsen (TQJ230) in lowering Lp(a) levels

CONTACTS AND LOCATIONS:
Locations (24):
- United States (24):
  - Parkway Medical Center, Birmingham, Alabama
  - National Heart Institute, Beverly Hills, California
  - Excel Medical Clinical Trials LLC, Boca Raton, Florida
  - Proactive Clinical Research, Fort Lauderdale, Florida
  - National Research Institute, Hialeah, Florida
  - Finlay Medical Research, Miami, Florida
  - Inpatient Research Clinical LLC, Miami Lakes, Florida
  - DBC Research USA, Pembroke Pines, Florida
  - Cardiology Partners Clinical Research Institute, Wellington, Florida
  - Cardiovascular Associates Research, Covington, Louisiana
  - Southern Clin Research Clinic, Zachary, Louisiana
  - Anderson Medical Research, Ft. Washington, Maryland
  - Capitol Cardiology Associates, Lanham, Maryland
  - Henry Ford Hospital, Detroit, Michigan
  - Aa Mrc Llc, Flint, Michigan
  - AB Clinical Trials, Las Vegas, Nevada
  - Clinical Research of South Nevada, Las Vegas, Nevada
  - Apex Cardiology Research Associates of Jackson, Jackson, Tennessee
  - North Hills Medical Research Inc, Bedford, Texas
  - Angiocardiac Care of Texas PA, Houston, Texas
  - Biopharma Informatic LLC, Houston, Texas
  - Clinical Trials of Texas, San Antonio, Texas
  - Javara Research, Alexandria, Virginia
  - Virginia Heart, Falls Church, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations. This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com.